CLINICAL TRIAL: NCT02288884
Title: The Use of a Silver Containing Dressing (Acticoat) on Wound Complication Rates Post Elective Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saskatchewan Health Authority - Regina Area (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RQhealth
Record Dates: First submitted 2014-11-07; First posted 2014-11-11 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-04

CONDITIONS: Surgical Wound Infection
Keywords: Complications; Cesarean Section; Wound; Infection (Following Delivery)
MeSH Terms: conditions — Surgical Wound Infection; Wounds and Injuries; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Silver containing dressing (Active Comparator): Subjects will have a silver containing dressing (Acticoat PostOp) applied at the time of elective cesarean section.
  Interventions: Device: Acticoat PostOp
- Standard dressing (Placebo Comparator): Subjects will have a standard dressing (OpSite PostOp) applied at the time of elective cesarean section.
  Interventions: Device: OpSite PostOp

INTERVENTIONS:
Device: Acticoat PostOp
  Arms: Silver containing dressing
Device: OpSite PostOp
  Arms: Standard dressing

SUMMARY:
The purpose of this study is to determine the effect of a silver containing dressing (Acticoat Post-Op) compared to a standard dressing (OpSite PostOp) on post elective cesarean section wound complications in obese women (BMI >35).

DETAILED DESCRIPTION:
Women scheduled for an elective cesarean section at term will be recruited to participate in this study. The investigators plan to recruit 100 women. Baseline demographic information will be obtained at the pre-op visit. Eligible subjects will be randomized to received a silver containing dressing (Acticoat PostOp) or the standard dressing (OpSite PostOp). A randomization table will be computer generated in blocks of 20. A sealed opaque envelope containing the assigned dressing will accompany the patient to the operating room. Standard antibiotic prophylaxis will be provided prior to skin incision. A subcuticular suture will be used for skin closure. At the time of skin closure, the envelope will be opened and the assigned dressing will be applied. The dressing will only be changed if it is saturated. The dressing will be removed at the time of discharge from hospital. A questionnaire regarding wound complications will be completed at the time of discharge from hospital, at 2 weeks post-op and 6 weeks post-op.

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for elective cesarean section
* BMI >35 at the pre-op visit
* consent to participate

Exclusion Criteria:

* allergy to silver
* immunocompromised (HIV/AIDS, on immunosuppressive medications)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Wound complication | 6 weeks post-op
  Composite of: wound infection treated with antibiotics, incision and drainage, wound requiring packing, or patient requiring medical attention for concerns about wound healing.

CONTACTS AND LOCATIONS:
Locations (1):
- Regina General Hospital, Regina, Saskatchewan, Canada